CLINICAL TRIAL: NCT06325553
Title: Incidence of Platelet Refractoriness in Adult Acute Leukemia Patients Receiving Prestorage-filtered Blood and Comparing With Historical Control
Brief Title: Incidence of Platelet Refractoriness in Adult Acute Leukemia Patients Receiving Prestorage Filtered Blood and Comparing With Historical Control
Acronym: PTR
Status: Recruiting | Type: Observational
Sponsor: Siriraj Hospital (Other)
Responsible Party: Principal Investigator, Weerapat Owattanapanich, Associate professor, Siriraj Hospital
Other Study IDs: 022_2566
Record Dates: First submitted 2024-03-15; First posted 2024-03-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Platelet Refractoriness in Adult Acute Leukemia
Keywords: Prestorage filtered blood; Platelet refractoriness in adult acute leukemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 1: Case group (PFB transfusion) Inclusion criteria
  1. Newly diagnosed acute leukemia (either acute myeloid leukemia (AML) or acute lymphoblastic leukemia (ALL) patients underwent intensive chemotherapy
  2. Age greater than 18 years
  3. Participants receiving an induction chemotherapy and at least one cycle of consolidation chemotherapy
  Exclusion criteria
  1. Participants with positive platelet antibody detected by SPRCA method at presentation
  Withdrawal or termination criteria
  1. Loss to follow up or death before completion of first consolidation chemotherapy
  2. Participants receiving granulocyte infusion during time of study
  3. Participants receiving SDP transfusion during time of study
- 2: Historical control group 1 (non-leukocyte depleted blood product) Inclusion criteria
  1. Newly diagnosed acute leukemia (either AML or ALL) patients underwent intensive chemotherapy during 2018-2022
  2. Age greater than 18 years
  3. Participants receiving an induction chemotherapy and at least one cycle of consolidation chemotherapy
  4. Participants receiving only non-leukocyte depleted blood products (LPB and LPPC)
  Exclusion criteria
  1. Loss to follow up or death before completion of first consolidation chemotherapy
  2. Participants receiving granulocyte infusion during time of study
- 3: Historical control group 2 (leukocyte depleted blood product) Inclusion criteria
  1. Newly diagnosed acute leukemia (either AML or ALL) patients underwent intensive chemotherapy during 2018-2022
  2. Age greater than 18 years
  3. Participants receiving an induction chemotherapy and at least one cycle of consolidation chemotherapy
  4. Participants receiving leukocyte depleted blood products (PFB and SDP)
  Exclusion criteria
  1. Loss to follow up or death before completion of first consolidation chemotherapy during 2018-2022
  2. Participants receiving granulocyte infusion during time of study
  3. Participants receiving non-leukocyte depleted blood products greater than 20% of all transfused blood products during induction and first consolidation chemotherapy

SUMMARY:
This research project is evaluate the incidence of platelet refractoriness in newly diagnosed acute leukemia patients receiving PFB during induction and first consolidation phase chemotherapy compared to 2 historical control groups which are patients receiving non-leukocyte depleted blood product group and leukocyte depleted blood product group and demonstrate cost-effectiveness of using blood products with filtered process to prevent clinical platelet refractoriness compare with using HLA-matched blood products after platelet refractoriness occurs

DETAILED DESCRIPTION:
This study the objective is to study and compare the incidence of Platelet Refractoriness. of the group that received PFB blood compared to the group that received LPPC/LPB blood in the past in patients with AML and ALL at Siriraj Hospital From the literature review, it was found that the incidence of Platelet Refractoriness of the group receiving LPPC/LPB blood in patients with AML and ALL was 46% and the incidence of Platelet Refractoriness Of the group receiving PFB blood in AML and ALL patients, it was 11% .But from the collection of blood bank data Siriraj Hospital during 2020-2021 found that the incidence of Platelet Refractoriness in AML and ALL patients who received PFB blood was approximately 27%. The researchers estimated that In this study There may be an incidence of Platelet Refractoriness. of the group receiving PFB blood in patients with AML and ALL was as high as 27%, and when determining the sample size in the group receiving LPPC/LPB blood, it was 2 times greater than the group receiving PFB blood and setting the standard value according to the table Z equal to 1.96 and The power of the test is 80% when the sample size is calculated with the formula Comparing the proportion values between two independent populations (Testing two independent proportion: Formula (without continuity correlation))

ELIGIBILITY:
Inclusion Criteria:

Case group (PFB transfusion) Inclusion criteria

1. Newly diagnosed acute leukemia (either acute myeloid leukemia (AML) or acute lymphoblastic leukemia (ALL) patients underwent intensive chemotherapy
2. Age greater than 18 years
3. Participants receiving an induction chemotherapy and at least one cycle of consolidation chemotherapy

Exclusion Criteria:

1. Participants with positive platelet antibody detected by SPRCA method at presentation

Historical control group 1 (non-leukocyte depleted blood product) Inclusion criteria 1.Newly diagnosed acute leukemia (either AML or ALL) patients underwent intensive chemotherapy during 2018-2022 2. Age greater than 18 years 3. Participants receiving an induction chemotherapy and at least one cycle of consolidation chemotherapy 4. Participants receiving only non-leukocyte depleted blood products (LPB and LPPC) Exclusion criteria

1. Loss to follow up or death before completion of first consolidation chemotherapy
2. Participants receiving granulocyte infusion during time of study

Historical control group 2 (leukocyte depleted blood product) Inclusion criteria

1. Newly diagnosed acute leukemia (either AML or ALL) patients underwent intensive chemotherapy during 2018-2022
2. Age greater than 18 years
3. Participants receiving an induction chemotherapy and at least one cycle of consolidation chemotherapy
4. Participants receiving leukocyte depleted blood products (PFB and SDP) Exclusion criteria

1. Loss to follow up or death before completion of first consolidation chemotherapy during 2018-2022 2. Participants receiving granulocyte infusion during time of study 3. Participants receiving non-leukocyte depleted blood products greater than 20% of all transfused blood products during induction and first consolidation chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient 18 years and older who were Newly diagnosed acute leukemia (either acute myeloid leukemia (AML) or acute lymphoblastic leukemia (ALL) patients underwent intensive chemotherapy
Sampling Method: Probability Sample
Enrollment: 252 (Estimated)
Dates: Start 2024-03-30 (Estimated); Primary Completion 2025-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Descriptive statistics | Through study completion and average of 1 year
  Qualitative variables (e.g. sex, underlying diseases) are presented as the frequency and percentage. Quantitative variables (e.g. age at diagnosis, follow-up time) are presented as mean and standard deviation if the data is normally distributed. Median and range are presented instead if the data is not normally distributed
Inferential statistics | Through study completion and average of 1 year
  The incidence of platelet refractoriness among each group are represented with percentage and associated 95% confidence interval (CI)

CONTACTS AND LOCATIONS:
Overall Officials: weerapat Owattanapanich, MD, Principal Investigator — Siriraj Hospital
Locations (1):
- Siriraj hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
IPD are available from the corresponding author on reasonable request
Supporting Information: Study Protocol